CLINICAL TRIAL: NCT02280213
Title: Comparison of Tracheal Intubation Using the Miller, Macintosh, Phillips and Wis-Hipple Blades During Infant Resuscitation: A Randomized Crossover Simulation Trial
Brief Title: Comparison Four Intubation Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/06
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation without chest compression (Experimental): Endotracheal intubation of infant mannikin using different laryngoscope blades (MAC, MIL, PHIL, WIS) during resuscitation without chest compressions.
  Interventions: Device: MIL; Device: MAC; Device: WIS; Device: PHIL
- Intubation with chest compression (Experimental): Endotracheal intubation of infant mannikin using different laryngoscope blades (MAC, MIL, PHIL, WIS) with uninterrupted chest compressions. Chest compressions with the two thumb-encircling hands technique were performed by the same Basic Life Support (BLS) instructor at a rate of 100 compressions per minute and at a depth of about 1.5 inches according to the European Resuscitation Council guidelines of 2010 year.
  Interventions: Device: MIL; Device: MAC; Device: WIS; Device: PHIL

INTERVENTIONS:
Device: MIL — Direct laryngoscopy 1
  Other Names: Miller blade
Device: MAC — Direct laryngoscopy 2
  Other Names: Macintosh blade
Device: WIS — Direct laryngoscopy 3
  Other Names: Wis-Hipple blade
Device: PHIL — Direct laryngoscopy 4
  Other Names: Phillips blade

SUMMARY:
Comparison of four laryngoscope blades (Miller, Macintosh, Phillips and Wis-Hipple) for infant intubation during resuscitation with and without chest compressions.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* paramedics
* no clinical experience in infant intubation

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to intubation | 1 day
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
Ease of Use | 1 day
  To access subjective opinions about the difficulty of the each intubation method, participants were asked to give a rating on a visual analogue scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult).
POGO score | 1 day
  The POGO score describes how much glottic opening is visible. A POGO score of 100% indicates visualization of the entire glottic opening from the anterior commissure of the vocal cords to the interarytenoid notch. A POGO score of 0% corresponds with no visualization of laryngeal structures.
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)
dental compression | 1 day
  pressure applied on the upper teeth (n=none, mild=1, moderate=2, severe=3)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland